CLINICAL TRIAL: NCT05221892
Title: Double Blind Evaluation of Gamma-aminobutyric Acid Tartarate 100 mg, Glutamic Acid 100 mg, Dibasic Calcium Phosphate 50 mg, Thiamine Nitrate 25 mg, Pyridoxine Chloride 10 mg and Cyanocobalamin 5 mcg Versus Ginger for Vertigo-kinetosis
Brief Title: Evaluation of Aminobutyric Acid, Glutamic Acid, Calcium, Thiamine, Pyridoxine and Cyanocobalamin as Therapy for Vertigo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, professor, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50635421.30000.5247
Record Dates: First submitted 2021-11-10; First posted 2022-02-03 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Vertigo
Keywords: vertigo; gamma aminobutyric acid; calcium; glutamic acid; thiamine; pyridoxine; cyanocobalamin; ginger
MeSH Terms: conditions — Vertigo | interventions — Glutamic Acid; calcium phosphate, dibasic, anhydrous; Thiamine; Vitamin B 12; ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test combination (Experimental): Gamma-aminobutyric acid tartrate 100mg, glutamic acid 100mg, dibasic calcium phosphate 50mg, thiamine nitrate 25mg, pyridoxine hydrochloride 10mg and cyanocobalamin 5mcg
  Interventions: Drug: Gamma-aminobutyric acid tartarate, glutamic acid, dibasic calcium phosphate, thiamine nitrate, pyridoxine chloride and cyanocobalamin
- Comparative medication (Active Comparator): Ginger extract 160mg (8mg gingerols)
  Interventions: Drug: Ginger

INTERVENTIONS:
Drug: Gamma-aminobutyric acid tartarate, glutamic acid, dibasic calcium phosphate, thiamine nitrate, pyridoxine chloride and cyanocobalamin — Tablets to be taken 30 minutes before each of 4 trips.
  Other Names: Gamma-aminobutyric acid tartarate, and combinations
  Arms: Test combination
Drug: Ginger — Tablets to be taken 30 minutes before each of 4 trips.
  Other Names: Zingiber officinale
  Arms: Comparative medication

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of a combination of aminobutyric acid, glutamic acid, calcium, thiamine, pyridoxine and cyanocobalamin as adjuvant therapy for vertigo comparatively to ginger under a double-blind randomized study design.

DETAILED DESCRIPTION:
Motion sickness is a chronic condition characterized by vestibular changes in response to stimuli caused either by movement or movement perception triggered by car, train, ship or aircraft transportation, amusement park rides, virtual reality and simulators, walking, exercising, as well as under the absence of gravity in space.The studied combination drug is composed by GABA (gamma-aminobutyric acid), the main inhibitory neurotransmitter of the central nervous system. The former lowers anxiety symptoms. Its precursor, glutamic acid, is the amino acid found in greater concentration under free form in the CNS; it is closely related to brain metabolism and, in contrast to GABA, it is the main excitatory neurotransmitter; glutamic acid also has anxyolytic therapeutic properties. Thiamine or vitamin B1 is a cofactor in the synthesis of acetylcholine, which plays a central role in the initiation and propagation of neural impulse in the CNS as well as it does in the skeletal and myocardial muscles. Pyridoxine or vitamin B6 plays a role in the synthesis of neurotransmitters such as dopamine as well as in the metabolism of tryptophan, resulting in an increase in serotonin so providing well-being and anxiety relief. Pyridoxine is essential for the proper functioning of the CNS (including at nausea and vomiting center). Cyancobalamin or Vitamin B12 plays a role in the growth and repair of nerve fibers. Importantly it also improves blood flow in the brain, with secondary vertigo improvement. The combined use of these substances provides relief of vertigo due to motion sickness. Zingiber officinale is a species of the Zingiberacaea family, widely used in traditional and herbal medicine for the treatment of various clinical conditions such as vertigo.

ELIGIBILITY:
Inclusion Criteria:

* clinical kinetosis
* female study subjects must agree in using contraceptives during study period
* dated informed consent read, understood and undersigned

Exclusion Criteria:

* hypersensitivity to the drugs of the study
* history of gallblader stones
* history of gastric mucosa inflammation
* arterial blood pressure >145/100 mmHg
* use of medication for kinetosis other than the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
motion sickness assessment questionnaire | 1 year
  The MSAQ consists of 16 questions, answered on a scale from one to nine points, which assesses the gastrointestinal, central and peripheral nervous system and soporous symptoms related to motion sickness.

CONTACTS AND LOCATIONS:
Overall Officials: carlos p nunes, MD, Principal Investigator — Fundação Educacional Serra dos Órgãos
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marx W, Ried K, McCarthy AL, Vitetta L, Sali A, McKavanagh D, Isenring L. Ginger-Mechanism of action in chemotherapy-induced nausea and vomiting: A review. Crit Rev Food Sci Nutr. 2017 Jan 2;57(1):141-146. doi: 10.1080/10408398.2013.865590. PMID 25848702
- [Background] Gianaros PJ, Muth ER, Mordkoff JT, Levine ME, Stern RM. A questionnaire for the assessment of the multiple dimensions of motion sickness. Aviat Space Environ Med. 2001 Feb;72(2):115-9. PMID 11211039
- [Background] Schmid R, Schick T, Steffen R, Tschopp A, Wilk T. Comparison of Seven Commonly Used Agents for Prophylaxis of Seasickness. J Travel Med. 1994 Dec 1;1(4):203-206. doi: 10.1111/j.1708-8305.1994.tb00596.x. PMID 9815340
- [Background] Surh Y. Molecular mechanisms of chemopreventive effects of selected dietary and medicinal phenolic substances. Mutat Res. 1999 Jul 16;428(1-2):305-27. doi: 10.1016/s1383-5742(99)00057-5. PMID 10518003
- [Background] Ali BH, Blunden G, Tanira MO, Nemmar A. Some phytochemical, pharmacological and toxicological properties of ginger (Zingiber officinale Roscoe): a review of recent research. Food Chem Toxicol. 2008 Feb;46(2):409-20. doi: 10.1016/j.fct.2007.09.085. Epub 2007 Sep 18. PMID 17950516
- [Background] Bailey-Shaw YA, Williams LA, Junor GA, Green CE, Hibbert SL, Salmon CN, Smith AM. Changes in the contents of oleoresin and pungent bioactive principles of Jamaican ginger (Zingiber officinale Roscoe.) during maturation. J Agric Food Chem. 2008 Jul 23;56(14):5564-71. doi: 10.1021/jf072782m. Epub 2008 Jun 20. PMID 18564850
- [Background] Calderon-Ospina CA, Nava-Mesa MO. B Vitamins in the nervous system: Current knowledge of the biochemical modes of action and synergies of thiamine, pyridoxine, and cobalamin. CNS Neurosci Ther. 2020 Jan;26(1):5-13. doi: 10.1111/cns.13207. Epub 2019 Sep 6. PMID 31490017
- [Background] Ezzat SM, Ezzat MI, Okba MM, Menze ET, Abdel-Naim AB. The hidden mechanism beyond ginger (Zingiber officinale Rosc.) potent in vivo and in vitro anti-inflammatory activity. J Ethnopharmacol. 2018 Mar 25;214:113-123. doi: 10.1016/j.jep.2017.12.019. Epub 2017 Dec 16. PMID 29253614
- [Background] Zempleni J, Suttie JW, Gregory JF III, Stover PJ. Handbook of Vitamins. Boca Raton, Florida, USA: CRC Press; 2013.
- [Result] Grontved A, Hentzer E. Vertigo-reducing effect of ginger root. A controlled clinical study. ORL J Otorhinolaryngol Relat Spec. 1986;48(5):282-6. doi: 10.1159/000275883. PMID 3537898
- [Result] Ernst E, Pittler MH. Efficacy of ginger for nausea and vomiting: a systematic review of randomized clinical trials. Br J Anaesth. 2000 Mar;84(3):367-71. doi: 10.1093/oxfordjournals.bja.a013442. PMID 10793599

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT05221892/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT05221892/SAP_001.pdf